CLINICAL TRIAL: NCT04567940
Title: ENRED@TE. Social Support in Southern Spain. Interventional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ENRED@TE
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Social Isolation
Keywords: Social isolation; Social support; Loneliness; Family support
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Behavioural multicomponent intervention
  Interventions: Behavioral: ENRED@TE: Behavioural multicomponent intervention
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: ENRED@TE: Behavioural multicomponent intervention — Information and awareness activities; activities for the acquisition of skills; activities that help the elderly to attend spaces for leisure, participation and maintenance and/or improvement of their personal relationships.
  Arms: Intervention group

SUMMARY:
The main objective to be achieved is to find out if the perceived social support, the perceived loneliness, the perceived social isolation and the family support of those over 65 years of age improve after participating in the Enréd@te project carried out by the Spanish Red Cross (CRE).

ELIGIBILITY:
Inclusion Criteria:

* People over 65 years
* Not institutionalised

Exclusion Criteria:

* Participants of other programs
* Difficulty responding to measurement scales due to language barriers
* Legal incapacitation
* People with a residence of less than 3 months in the city

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Social isolation | 6 months
  Duke-UNC Functional Social Support Questionnaire (Bellón et al. 1996) is an eight-item instrument to measure the strength of the person's social support network. Each item is ranged from 1 to 5 points, where high scores represent greater social support.
Loneliness | 6 months
  UCLA Loneliness Scale (Russell DW, 1996) which is a 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. This tool use a 4-point rating scale (1= never; 4 = always). High values mean more loneliness.

SECONDARY OUTCOMES:
Detection of risk situations or social problems | 6 months
  Gijón socio-family assessment scale (García González et al. 1999) allows the detection of risk situations or social problems. Values range from 3 to 15. Higher values mean more severe social decline.

CONTACTS AND LOCATIONS:
Locations (1):
- Maimónides Biomedical Research Institute of Córdoba, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: No